CLINICAL TRIAL: NCT06809075
Title: Immunological Reset to Allow Access to HLA Compatible Transplantation in Highly Sensitized Kidney Transplant Candidates Through Non-myeloablative Autologous Stemm Cell Transplantation (RESET TRIAL)
Brief Title: Immunological Reset to Allow Access to HLA Compatible Transplantation in Highly Sensitized Kidney Transplant Candidates Through Non-myeloablative Autologous Stemm Cell Transplantation
Acronym: RESET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RESET; 2023-506478-11-01 (EU CTIS Number)
Record Dates: First submitted 2024-10-03; First posted 2025-02-05 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Kidney Disease; Kidney Transplant; Kidney Transplant Candidates
Keywords: HLA; TPHa; Kidney transplant; hypersensitized patient; cPRA; immunosuppression; DSA; aHSCT
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- hypersensitive patients undergoing aHSCT (Experimental): hypersensitive patients undergoing aHSCT. All patients in this study participate in this arm.
  Interventions: Procedure: hematopoietic precursor transplantation (TPHa)

INTERVENTIONS:
Procedure: hematopoietic precursor transplantation (TPHa) — An apheresis is performed on the patients and a selection of CD34 hematopoietic progenitors is performed. Subsequently, conditioning is performed with cyclophosphamide, thymoglobulin, corticosteroids and rituximab to subsequently infuse the hematopoietic precursors.

SUMMARY:
This is a study for hypersensitized patients who have been waiting for more than 3 years for an offer for a kidney transplant. The objective is to perform a transplant of autologous hematopoietic precursors with the aim of producing what we call an immunological reset to make the maximum number of anti-HLA antibodies disappear and thus increase the chances of the patient receiving an offer for a kidney transplant.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be able to understand and give written consent.
2. Women and men between 18 and 65 years old.
3. Patients with chronic kidney disease who are on renal therapy replacement with dialysis.
4. Patient who is on the waiting list for kidney transplant from a death donor and who has not received an offer for a compatible transplant in the last 3 years within the national PATHI prioritization program.
5. cPRA calculated of more than 97% and having been in the program of prioritization for more than 3 years
6. Positive IgG serologies for Cytomegalovirus and Epstein Barr.
7. Women of childbearing potential must have a negative pregnancy test upon entry to the study and must agree to use safe contraceptive methods according to the guideline CTFG recommendations on contraception in clinical trials during duration of the study (condoms are considered safe methods male and female, oral contraceptives, etc.).
8. Patients vaccinated against tetanus, influenza, pneumococcus and herpes zoster

Exclusion Criteria:

1. Current known infection, recurrent bacteria, virus, fungus or fungus bacteria, or other infections (such as HIV, hepatitis B, hepatitis C, or zoster).
2. Concomitant serious uncontrolled major organ disease.
3. Any infection that requires hospitalization and intravenous treatment with antibiotics during the 4 weeks prior to screening, or oral treatment with antibiotics the previous 2 weeks.
4. Patients with primary or secondary immunodeficiencies.
5. Patient with an active history of tuberculosis (even if treated) or patients with untreated latent tuberculosis.
6. Malignancy during the 5 years prior to screening, except for carcinoma of the basal cell or squamous cell carcinoma properly removed.
7. Known abuse of alcohol, drugs or chemicals within 1 year prior to screening.
8. Patients with complicated peripheral venous access
9. Neutropenia (ANC <1000/uL) or thrombocytopenia (platelet count <100,000/uL) during the 4 weeks prior to screening.
10. Severe allergic or anaphylactic reactions to human monoclonal antibodies, humanized or murine.
11. Treatment with any investigational agent during the 4 weeks (or 5 half-lives of the investigational drug, whichever is longer) prior to screening.
12. Immunization with live vaccine during the 2 months prior to screening.
13. Pregnant or breastfeeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the impact of autologous hematopoietic stem cell transplantation (aHSCT) | from enrolment to 12 months post-TPHa
  Variable composed with the proportion of patients in whom ≥10 HLA, class I or class II antibodies are eliminated (undetectable or <1000 MFI) or the percentage of baseline cPRA is decreased at 6 months after aHSCT, in the absence of severe undesirable effects related to the treatment.
Proportion of patients achieving all of the following items at 6 months post-aHSCT or at the time of kidney transplant, if a compatible offer is received | from enrolment to 12 months post-aHSCT
  Proportion of patients achieving all of the following items at 6 months post-aHSCT or at the time of kidney transplant, if a compatible offer is received
  * Elimination/reduction of HLA antibody-secreting plasma cells in the bone marrow
  * Absence/reduction of HLA-specific memory B cells in circulation

SECONDARY OUTCOMES:
Total number of HLA antibodies eliminated | from enrolment to 6 months post-aHSCT
  Total number of HLA antibodies eliminated
Average number of HLA antibodies eliminated | from enrolment to 6 months post-aHSCT
  Average number of HLA antibodies eliminated
Mean reduction in MFI of immunodominant HLA antibody, class I and class II | from enrolment to 6 months post-aHSCT
  Mean reduction in MFI of immunodominant HLA antibody, class I and class II
Proportion of patients transplanted with a compatible donor | from enrolment to 12 months post-aHSCT
  Proportion of patients transplanted with a compatible donor
Adverse reactions related to aHSCT | from enrolment to 12 months post-aHSCT
  Mesure the number of adverse reactions related to aHSCT
Incidence of opportunistic infections | From aHSCT to 12 months after aHSCT or 12 months after kidney transplant (if it's occurs)
  Mesure the Incidence of opportunistic infections in treated patients
Incidence of clinical and/or subclinical rejection mediated by antibodies in the first year after kidney transplantation | from kidney trasplantation to 12 months after
  Incidence of clinical and/or subclinical rejection mediated by antibodies in the first year after kidney transplantation
Proportion of patients free of DSA and/or donor-specific memory B cells at 1 year after kidney transplant | from kidney transplant to 1 year post kidney transplant
  Proportion of patients free of DSA and/or donor-specific memory B cells at 1 year after kidney transplant
Changes in the clonal and phenotypic repertoire of B and T cells. | From aHSCT to 12 months after aHSCT or 12 months after kidney transplant (if it's occurs)
  Changes in the clonal and phenotypic repertoire of B and T cells mesure with cytometry

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided